CLINICAL TRIAL: NCT02730663
Title: A Prospective, Multi-center, Single Arm, Non-inferiority, Open-label, Pivotal Study to Evaluate the Effectiveness and Safety of EUS -Guided Transluminal Drainage With 'Niti-S SPAXUS Stent' for the Treatment of Pancreatic Pseudocyst
Brief Title: A Study to Evaluate the Effectiveness and Safety of EUS-guided Transluminal Drainage With 'Niti-S SPAXUS Stent'
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taewoong Medical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPAXUS-001
Record Dates: First submitted 2016-03-28; First posted 2016-04-06 (Estimated); Results first posted 2019-07-01 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-04

CONDITIONS: Pancreatic Pseudocyst
Keywords: Endoscopic ultrasound guided transluminal drainage
MeSH Terms: conditions — Pancreatic Pseudocyst

STUDY DESIGN:
Intervention Model Description: The investigational device (ID) 'Niti-S SPAXUS Stent' is used for drainage of cystic fluid by being connected to the pancreatic pseudocyst through human organs such as stomach or duodenum. It is composed with a stent made of nitinol and introducer system.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Niti-S SPAXUS Stent (Experimental): Niti-S SPAXUS Stent (TaeWoong Medical Co., Ltd. Korea)
  Interventions: Device: Niti-S SPAXUS Stent

INTERVENTIONS:
Device: Niti-S SPAXUS Stent — Endoscopic Ultrasound-Guided Transluminal drainage

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of endoscopic ultrasound (EUS)-guided transluminal drainage with 'Niti-S SPAXUS Stent' for the treatment of pancreatic pseudocyst.

DETAILED DESCRIPTION:
'Niti-S SPAXUS Stent' is a newly designed lumen-apposing fully covered self-expandable metal stent. It is indicated for use in patients with pancreatic pseudocyst. Consecutive subject data should be collected at discharge, stent removal (day 30 or 60), and day 20 post Niti-S SPAXUS stent removal.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic pseudocyst ≥6cm in size, with ≥70% fluid content that is eligible for transluminal drainage
* Patient willing to provide written informed consent and comply with follow-up requirements

Exclusion Criteria:

* Ineligible for endoscopic intervention
* Pancreatic pseudocyst with severe internal septation
* Platelet count < 60,000 cells/mm3 or international normalized ratio (INR) >1.5
* Hemodynamic instability (e.g. shock)
* Active infectious disease (e.g. endocarditis, meningitis)
* Participating in any other investigational drug or device clinical trial within past 3 months
* Female of child-bearing potential who are unable to take adequate contraceptive precautions, are known to be pregnant, or are currently breastfeeding an infant

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-03-21 (Actual); Primary Completion 2017-06-14 (Actual); Study Completion 2017-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jong Ho Moon, PhD, MD, Principal Investigator — Soon Chun Hyang University; Sang Soo Lee, PhD, MD, Principal Investigator — Asan Medical Center; Jong Kyun Lee, PhD, MD, Principal Investigator — Samsung Medical Center; Seung-Ok Lee, PhD, MD, Principal Investigator — Chonbuk National University Hospital; Chang Min Cho, PhD, MD, Principal Investigator — Kyungpook National University Medical Center; Se Woo Park, PhD, MD, Principal Investigator — Hallym University Dongtan Sacred Heart Hospital
Locations (6):
- South Korea (6):
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si, Gyeonggi-do
  - Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si, Gyeonggi-do
  - Kyungpook National University Medical Center, Daegu
  - Chonbook National University Hospital, Jeonju
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No
Oct, 2016

REFERENCES:
- [Derived] Song TJ, Lee SS, Moon JH, Choi HJ, Cho CM, Lee KH, Park SW, Kim SH, Lee SO, Lee YN, Lee JK. Efficacy of a novel lumen-apposing metal stent for the treatment of symptomatic pancreatic pseudocysts (with video). Gastrointest Endosc. 2019 Sep;90(3):507-513. doi: 10.1016/j.gie.2019.05.033. Epub 2019 May 30. PMID 31152738

RESULTS

PARTICIPANT FLOW:
Recruitment Details: It took about 15 months from the approval of the Ministry of Food and Drug Safety(MFDS) and the IRB, including the subject enrollment period of about 13 months and the follow-up period of 2 months at maximum.
Period: Overall Study
Arm/Group | Niti-S SPAXUS Stent
Started (1 subject in screening failure(impossible to undergo the stent procedure)) | 36
Completed | 35
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Niti-S SPAXUS Stent
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.51 (13.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Korea | 35
Height [Mean (Inter-Quartile Range); unit: cm] | 167.82 [144.30 to 182.30]
Body weight [Mean (Inter-Quartile Range); unit: kg] | 64.34 [43.50 to 96.00]
History of smoking [Number; unit: participants]
  Current Smoker | 13
  Ex-Smoker | 10
  Non-Smoker | 12
Alcohol drinking [Number; unit: participants]
  Current Drinker | 13
  Ex-Drinker | 14
  Non-Drinker | 8
History of allergy [Number; unit: participants]
  Yes | 2
  No | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Success
Description: Clinical success is defined as ≥50% decrease in pancreatic pseudocyst size measured on Computed Tomography (CT)
Time Frame: at stent removal (Day 30 or Day 60)
Population: The analysis is performed in the subjects who underwent the Niti-S SPAXUS stent and have the results of effectiveness assessment at the time point of the stent removal among those who satisfy the inclusion • exclusion criteria, consented to participate in the study
Measure: Number; unit: participants
Arm/Group | Niti-S SPAXUS Stent
Number analyzed (Participants) | 34
participants | 33
Statistical Analysis 1: Comparison: Niti-S SPAXUS Stent; The clinical success rate at the time point of stent removal is reported 86.2% according to the approval data of the commercially available AXIOS stent submitted to the US FDA. The clinical success rates of EUS-guided transluminal drainage using a lumen-appending stent were 93.3% (29 cases), 100% (8 cases) and 100% (7 cases) respectively in the studies performed afterwards by Shah RJ (2015), Gornals JB (2012) and Moon JH (2014). The weighted average calculated for each study was about 96%; Test type: Non-Inferiority — The number and percentage of patients who achieved clinical success at the time of stent removal are presented. A one-sided 97.5% confidence interval is to be calculated to confirm the degree of non-inferiority for the reference value (96%) and the difference (Investigational device - reference value) and if the lower limit of the confidence interval is -10% or higher, the noninferiority will be considered to be confirmed; p = 0.05, t-test, 2 sided — A two-tail test was performed for statistics at a significance level of 0.05 unless otherwise specified; Reference value = -0.07

2. Secondary Outcome: Number of Participants With Technical Success
Description: Technical success is defined as successful placement of the Niti-S SPAXUS stent across the gastric(or duodenal) wall to the pseudocyst with visualization of the pseudocyst fluid drainage through the stent by endoscopy.
Time Frame: Day 1
Population: If the stent is deployed successfully in the gastrointestinal tract and the pseudocyst, and if the drainage is confirmed visually, it is considered technically successful
Measure: Count of Participants; unit: Participants
Arm/Group | Niti-S SPAXUS Stent
Number analyzed (Participants) | 34
Participants | 33

3. Secondary Outcome: Number of Participants With Stent Lumen Patency
Description: Stent lumen patency will be evaluated by endoscopy.
Time Frame: up to 60 days (at stent removal, Day 30 or 60)
Population: The stent lumen patency will be evaluated by the investigator at Day 30 or 60 (± 10 days) after the procedure of the Niti-S SPAXUS stent through clinical symptoms and endoscopy.
Measure: Count of Participants; unit: Participants
Arm/Group | Niti-S SPAXUS Stent
Number analyzed (Participants) | 34
Participants | 34

4. Secondary Outcome: Number of Participants With Stent Removal Success
Description: Stent removal success is defined as successful removal of the Niti-S SPAXUS stent using a standard endoscopic forceps or snare.
Time Frame: up to 60 days (at stent removal, Day 30 or 60)
Population: When the Niti-S SPAXUSTM Stent is successfully removed by using forceps or snare through endoscopy as the treatment is succeeded clinically at Day 30 or 60 (± 10 days) according to standard procedures and the criteria for stent removal are met, it is considered as the stent removal success.
Measure: Count of Participants; unit: Participants
Arm/Group | Niti-S SPAXUS Stent
Number analyzed (Participants) | 34
Participants | 34

5. Secondary Outcome: Procedure Time
Description: Procedure time is measured as time from insertion until removal of endoscope. Procedure time 1: The time from the moment that the endoscope is inserted into the oral cavity to the time point at which the endoscope is removed. (sec) Procedure time 2: The time from the puncture time to the point at which the ultrasound endoscope was removed. (sec)
Time Frame: 1 day
Population: The time is measured from the moment that the endoscope is inserted into the oral cavity to the time point at which the endoscope is removed.
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Niti-S SPAXUS Stent
Number analyzed (Participants) | 34
sec
  Procedure time 1 | 1074.88 (618.30)
  Procedure time 2 | 618.12 (341.63)

6. Secondary Outcome: Number of Participants With Procedural/Device Related Serious Adverse Events
Description: The incidence of serious adverse events related to the procedure or the Niti-S SPAXUSTM stent is assessed at Day 20 after the stent removal
Time Frame: up to 90 days (at Day 20 post stent removal)
Population: * Resulted in death or life threatening
    * Required inpatient hospitalization or prolongation of existing hospitalization ③ Resulted in persistent or significant disability/incapacity ④ Caused a congenital anomaly/birth defect
Measure: Number; unit: participants
Arm/Group | Niti-S SPAXUS Stent
Number analyzed (Participants) | 35
participants | 14

7. Secondary Outcome: Other Adverse Events
Description: The severity and incidence of all other adverse events than those mentioned above occurred during the follow-up period were evaluated at Day 20 day after the stent removal.
Time Frame: up to 90 days (at Day 20 post stent removal)
Population: The severity and incidence of all other adverse events than those mentioned above occurred during the follow-up period were evaluated at Day 20 day after the stent removal.
Measure: Number; unit: case
Arm/Group | Niti-S SPAXUS Stent
Number analyzed (Participants) | 35
case | 154

ADVERSE EVENTS:
Time Frame: 3months
Description: An "Adverse Event (AE)" refers to any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device.
  Serious Adverse Event /Adverse Device Effect refers to the adverse events or adverse device effects occurred due to the investigational device, which is applicable to any of the consequences.
Arm/Group | Niti-S SPAXUS Stent
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 14/35
Other Adverse Events (participants affected / at risk) | 29/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Niti-S SPAXUS Stent (N=35)
Upper gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1)
Aggravated Walled off necrosis (Gastrointestinal disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Peripancreatic abscess (Infections and infestations) | 1 (1)
Pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Abdominal pain (LUQ pain) -> wall-off necrosis (Gastrointestinal disorders) | 1 (1)
Infected pseudocyst (Infections and infestations) | 3 (3)
Cerebral infarction (Nervous system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Necrotizing pseudocyst (Gastrointestinal disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Niti-S SPAXUS Stent (N=35)
Abdominal pain etc. (Gastrointestinal disorders) | 24 (69)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (1)
Pyrexia etc. (General disorders) | 17 (23)
Cholelithiasis etc. (Hepatobiliary disorders) | 2 (2)
Pancreas infection etc. (Infections and infestations) | 7 (7)
Pancreatic leak (Injury, poisoning and procedural complications) | 1 (1)
Blood pressure decreased (Investigations) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 9 (12)
Flank pain (Musculoskeletal and connective tissue disorders) | 6 (7)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-08): https://cdn.clinicaltrials.gov/large-docs/63/NCT02730663/Prot_SAP_000.pdf